CLINICAL TRIAL: NCT03651765
Title: Long Term Extension Trial of Setmelanotide (RM-493) for Patients Who Have Completed a Trial of Setmelanotide for the Treatment of Obesity Associated With Genetic Defects Upstream of the MC4 Receptor in the Leptin-melanocortin Pathway
Brief Title: Long Term Extension Trial of Setmelanotide
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-022; 2017-005006-35 (EudraCT Number)
Record Dates: First submitted 2018-01-18; First posted 2018-08-29 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Obesity Associated With Defects in Leptin-melanocortin Pathway
Keywords: setmelanotide; RM-493; obesity; leptin-melanocortin; melanocortin 4 receptor
MeSH Terms: conditions — Obesity | interventions — setmelanotide

STUDY DESIGN:
Intervention Model Description: Open label treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setmelanotide (Experimental): Participants received setmelanotide at the same starting dose as received in the index trials as a Subcutaneous (SC) injection once daily for up to 5.6 years in this extension trial.
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — Once daily subcutaneous injection
  Other Names: RM-493

SUMMARY:
This was a long-term extension trial to study the safety and tolerability of continued setmelanotide treatment in participants who had completed a previous clinical trial on treatment with setmelanotide for obesity associated with genetic defects upstream of the Melanocortin-4 (MC4) receptor in the leptin-melanocortin pathway.

DETAILED DESCRIPTION:
The primary objectives of this extension trial were to explore the long-term safety and tolerability of setmelanotide for up to 7 years or until drug was otherwise available through authorized use. Participants entered this protocol immediately upon completion of their index protocol such that dosing of setmelanotide continued without gaps in therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants aged 2 or older (or aged >2 years as per local regulations) who had completed participation in a previous setmelanotide trial and demonstrated adequate safety and meaningful clinical benefit (efficacy)
2. Participant and/or parent or guardian was able to communicate with the investigator, understand and sign the written informed consent/assent, and comply with the trial requirements
3. Agree to use a highly effective form of contraception throughout the trial

Key Exclusion Criteria:

1. Pregnant and/or breastfeeding women
2. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions (excluding non-invasive basal or squamous cell lesion)
3. Current, clinically significant disease
4. Documented diagnosis of schizophrenia, bipolar disorder, personality disorder, major depressive disorder, or other psychiatric disorder(s)
5. Suicidal ideation, attempt or behavior
6. History of significant liver disease
7. Moderate to severe renal dysfunction as defined by a glomerular filtration rate (GFR)<30 milliliters per minute (mL/min).
8. History or close family history of melanoma or participant history of oculocutaneous albinism

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (27):
- United States (15):
  - Synexus Clinical Research US, Inc. - Phoenix Southeast, Chandler, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - San Diego Wake Research, San Diego, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Baystate Medical Center, Springfield, Massachusetts
  - University at Buffalo, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research, Raleigh, North Carolina
  - Obesity Institute, Geisinger Clinic, Danville, Pennsylvania
  - Childrens Hospital of Philadephia, Philadelphia, Pennsylvania
  - Synexus Clinical Research US, Inc.- Primary Care Associates, PC, Anderson, South Carolina
  - Wake Research TN, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Seattle Children's Research Institute, Seattle, Washington
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin
- University of Alberta, Edmonton, Alberta, Canada
- France (2):
  - Hôpital Trousseau, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University of Leipzig, Leipzig
  - University of Ulm, Ulm
- University General Hospital of Patras, Rio, Greece
- Erasmus MC, Rotterdam, Netherlands
- Universidad Autónoma de Madrid, Madrid, Spain
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Wellcome Trust-MRC Institute of Metabolic Science, Cambridge
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth CL, Scimia C, Shoemaker AH, Gottschalk M, Miller J, Yuan G, Malhotra S, Abuzzahab MJ. Setmelanotide for the treatment of acquired hypothalamic obesity: a phase 2, open-label, multicentre trial. Lancet Diabetes Endocrinol. 2024 Jun;12(6):380-389. doi: 10.1016/S2213-8587(24)00087-1. Epub 2024 Apr 30. PMID 38697184
- [Derived] Meyer JR, Krentz AD, Berg RL, Richardson JG, Pomeroy J, Hebbring SJ, Haws RM. Kidney failure in Bardet-Biedl syndrome. Clin Genet. 2022 Apr;101(4):429-441. doi: 10.1111/cge.14119. PMID 35112343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from previous index trials (RM-493-011[NCT02507492], RM-493-012 [NCT02896192], RM-493-014[NCT03013543], RM-493-015 [NCT03287960], RM-493-023 [NCT03746522], RM-493-030 [NCT04725240], RM-493-034 [NCT04963231] with rare genetic, syndromic, or acquired diseases of obesity upstream of the Melanocortin-4 receptor (MC4R) in the melanocortin-leptin pathway and other abnormalities of the MC4R pathway and wished to continue with setmelanotide treatment were enrolled in this extension trial.
Pre-assignment Details: A total of 205 participants were enrolled in the study.
Period: Overall Study
Arm/Group | Setmelanotide
Started | 205
Completed | 89
Not Completed | 116
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 18
Not completed — Lost to Follow-up | 5
Not completed — Non-Compliance with Study Drug | 4
Not completed — Physician Decision | 6
Not completed — Pregnancy | 1
Not completed — Discontinued by Sponsor | 40
Not completed — Withdrawal by Parent/Guardian | 6
Not completed — Withdrawal by Subject | 24
Not completed — Miscellaneous | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all participants who received at least one dose of received at least 1 dose of setmelanotide in this extension trial.
Groups:
- Setmelanotide: Participants received setmelanotide at the same starting dose as received in the index trials as a SC injection once daily for up to 5.6 years in this extension trial.
Arm/Group | Setmelanotide
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.7 (14.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 167
  More than one race | 0
  Unknown or Not Reported | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 171
  Unknown or Not Reported | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE was defined as any AE that began or worsened in intensity on or after the date of the first administration of study drug.
Time Frame: From first dose up to 5.6 years
Population: SAS included all participants who received at least one dose of received at least 1 dose of setmelanotide in this extension trial.
Measure: Number; unit: Participants
Arm/Group | Setmelanotide
Number analyzed (Participants) | 205
Participants | 198

ADVERSE EVENTS:
Time Frame: From first dose up to 5.6 years
Description: SAS included all participants who received at least one dose of received at least 1 dose of setmelanotide in this extension trial.
Arm/Group | Setmelanotide
All-Cause Mortality (participants affected / at risk) | 0/205
Serious Adverse Events (participants affected / at risk) | 27/205
Other Adverse Events (participants affected / at risk) | 198/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide (N=205)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 1
Pilonidal disease (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Suicidal ideation (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 3
Seizure (Nervous system disorders) | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Muscle spasticity (Nervous system disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Angle closure glaucoma (Eye disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Setmelanotide (N=205)
Nasopharyngitis (Infections and infestations) | 32
Upper Respiratory Tract Infection (Infections and infestations) | 36
Covid-19 (Infections and infestations) | 60
Influenza (Infections and infestations) | 22
Urinary Tract Infection (Infections and infestations) | 17
Gastroenteritis (Infections and infestations) | 15
Ear Infection (Infections and infestations) | 12
Bronchitis (Infections and infestations) | 8
Gastroenteritis Viral (Infections and infestations) | 7
Viral Upper Respiratory Tract Infection (Infections and infestations) | 9
Otitis Media (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 7
Fungal Infection (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 7
Laryngitis (Infections and infestations) | 4
Oral Candidiasis (Infections and infestations) | 3
Paronychia (Infections and infestations) | 4
Pharyngitis Streptococcal (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 3
Respiratory Tract Infection (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 3
Subcutaneous Abscess (Infections and infestations) | 3
Viral Infection (Infections and infestations) | 4
Body Tinea (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 3
Lower Respiratory Tract Infection (Infections and infestations) | 3
Onychomycosis (Infections and infestations) | 3
Postoperative Wound Infection (Infections and infestations) | 2
Tinea Versicolour (Infections and infestations) | 3
Tooth Abscess (Infections and infestations) | 3
Tooth Infection (Infections and infestations) | 3
Vulvovaginal Candidiasis (Infections and infestations) | 2
Abscess Limb (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 2
Furuncle (Infections and infestations) | 2
Gastrointestinal Candidiasis (Infections and infestations) | 1
Gastrointestinal Infection (Infections and infestations) | 2
Gastrointestinal Viral Infection (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 2
Implant Site Infection (Infections and infestations) | 1
Oesophageal Candidiasis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 2
Otitis Externa (Infections and infestations) | 2
Otitis Externa Fungal (Infections and infestations) | 1
Pilonidal Disease (Infections and infestations) | 1
Pulpitis Dental (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 2
Acute Sinusitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bacterial Vaginosis (Infections and infestations) | 1
Carbuncle (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Eye Infection (Infections and infestations) | 1
Gastrointestinal Fungal Infection (Infections and infestations) | 1
Genital Candidiasis (Infections and infestations) | 1
Genital Herpes (Infections and infestations) | 1
Groin Abscess (Infections and infestations) | 1
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1
Herpes Simplex (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infected Bite (Infections and infestations) | 1
Injection Site Abscess (Infections and infestations) | 1
Injection Site Cellulitis (Infections and infestations) | 1
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 1
Ludwig Angina (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Otitis Media Acute (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pericoronitis (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Post-Acute Covid-19 Syndrome (Infections and infestations) | 1
Pustule (Infections and infestations) | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 1
Retinitis (Infections and infestations) | 1
Skin Bacterial Infection (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Streptococcal Infection (Infections and infestations) | 1
Systemic Viral Infection (Infections and infestations) | 1
Tinea Pedis (Infections and infestations) | 1
Tonsillitis Streptococcal (Infections and infestations) | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 110
Acanthosis Nigricans (Skin and subcutaneous tissue disorders) | 10
Acne (Skin and subcutaneous tissue disorders) | 11
Eczema (Skin and subcutaneous tissue disorders) | 11
Skin Depigmentation (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Hidradenitis (Skin and subcutaneous tissue disorders) | 7
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 5
Melanoderma (Skin and subcutaneous tissue disorders) | 6
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 6
Papule (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 5
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 5
Skin Lesion (Skin and subcutaneous tissue disorders) | 4
Alopecia Areata (Skin and subcutaneous tissue disorders) | 2
Cafe Au Lait Spots (Skin and subcutaneous tissue disorders) | 4
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4
Vitiligo (Skin and subcutaneous tissue disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 3
Erythema Ab Igne (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 2
Nail Discolouration (Skin and subcutaneous tissue disorders) | 2
Perioral Dermatitis (Skin and subcutaneous tissue disorders) | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 2
Seborrhoea (Skin and subcutaneous tissue disorders) | 2
Skin Striae (Skin and subcutaneous tissue disorders) | 2
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1
Ephelides (Skin and subcutaneous tissue disorders) | 1
Erythema Annulare (Skin and subcutaneous tissue disorders) | 1
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1
Keloid Scar (Skin and subcutaneous tissue disorders) | 1
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1
Lichenification (Skin and subcutaneous tissue disorders) | 1
Nail Disorder (Skin and subcutaneous tissue disorders) | 1
Nail Ridging (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 1
Skin Wrinkling (Skin and subcutaneous tissue disorders) | 1
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1
Injection Site Erythema (General disorders) | 43
Injection Site Induration (General disorders) | 35
Injection Site Pruritus (General disorders) | 38
Fatigue (General disorders) | 22
Injection Site Pain (General disorders) | 26
Injection Site Bruising (General disorders) | 25
Injection Site Oedema (General disorders) | 16
Pyrexia (General disorders) | 15
Injection Site Haemorrhage (General disorders) | 12
Oedema Peripheral (General disorders) | 7
Injection Site Haematoma (General disorders) | 5
Injection Site Reaction (General disorders) | 6
Non-Cardiac Chest Pain (General disorders) | 5
Injection Site Discolouration (General disorders) | 5
Asthenia (General disorders) | 4
Influenza Like Illness (General disorders) | 4
Illness (General disorders) | 1
Pain (General disorders) | 3
Application Site Erythema (General disorders) | 1
Chest Pain (General disorders) | 2
Feeling Cold (General disorders) | 2
Gait Disturbance (General disorders) | 2
Hangover (General disorders) | 1
Inflammation (General disorders) | 1
Injection Site Irritation (General disorders) | 2
Chills (General disorders) | 1
Complication Associated With Device (General disorders) | 1
Fat Tissue Increased (General disorders) | 1
Generalised Oedema (General disorders) | 1
Injection Site Discharge (General disorders) | 1
Injection Site Granuloma (General disorders) | 1
Injection Site Hypertrophy (General disorders) | 1
Injection Site Mass (General disorders) | 1
Injection Site Swelling (General disorders) | 1
Injection Site Urticaria (General disorders) | 1
Malaise (General disorders) | 1
Medical Device Site Haemorrhage (General disorders) | 1
Medical Device Site Pain (General disorders) | 1
Oedema (General disorders) | 1
Vessel Puncture Site Haematoma (General disorders) | 1
Nausea (Gastrointestinal disorders) | 28
Abdominal Pain Upper (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 21
Diarrhoea (Gastrointestinal disorders) | 17
Abdominal Pain (Gastrointestinal disorders) | 20
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 10
Tongue Pigmentation (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Oral Pigmentation (Gastrointestinal disorders) | 5
Abdominal Distension (Gastrointestinal disorders) | 4
Gingival Hyperpigmentation (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Abdominal Discomfort (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 2
Food Poisoning (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gingival Recession (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Tooth Impacted (Gastrointestinal disorders) | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Anal Fissure (Gastrointestinal disorders) | 1
Dental Caries (Gastrointestinal disorders) | 1
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 1
Gastrointestinal Tract Mucosal Pigmentation (Gastrointestinal disorders) | 1
Gingival Discolouration (Gastrointestinal disorders) | 1
Gingival Pain (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1
Lip Dry (Gastrointestinal disorders) | 1
Lymphoid Hyperplasia Of Intestine (Gastrointestinal disorders) | 1
Mouth Ulceration (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oesophageal Spasm (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral Lichen Planus (Gastrointestinal disorders) | 1
Periodontal Disease (Gastrointestinal disorders) | 1
Rectal Discharge (Gastrointestinal disorders) | 1
Swollen Tongue (Gastrointestinal disorders) | 1
Tongue Coated (Gastrointestinal disorders) | 1
Tongue Discolouration (Gastrointestinal disorders) | 1
Tooth Erosion (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 60
Dizziness (Nervous system disorders) | 16
Migraine (Nervous system disorders) | 9
Seizure (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 4
Disturbance In Attention (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 3
Dizziness Postural (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Restless Legs Syndrome (Nervous system disorders) | 1
Sinus Headache (Nervous system disorders) | 2
Sleep Paralysis (Nervous system disorders) | 1
Altered State Of Consciousness (Nervous system disorders) | 1
Bell's Palsy (Nervous system disorders) | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 1
Cerebrospinal Fluid Leakage (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Facial Paralysis (Nervous system disorders) | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1
Nerve Compression (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Occipital Neuralgia (Nervous system disorders) | 1
Ophthalmic Migraine (Nervous system disorders) | 1
Parosmia (Nervous system disorders) | 1
Peroneal Nerve Palsy (Nervous system disorders) | 1
Petit Mal Epilepsy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Taste Disorder (Nervous system disorders) | 1
Tension Headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 13
Blood Creatine Phosphokinase Increased (Investigations) | 11
Gamma-Glutamyltransferase Increased (Investigations) | 7
Glycosylated Haemoglobin Increased (Investigations) | 6
Blood Cholesterol Increased (Investigations) | 6
Blood Triglycerides Increased (Investigations) | 5
C-Reactive Protein Increased (Investigations) | 5
Hepatic Enzyme Increased (Investigations) | 5
Low Density Lipoprotein Increased (Investigations) | 5
Aspartate Aminotransferase Increased (Investigations) | 4
Blood Bilirubin Increased (Investigations) | 4
Blood Lactate Dehydrogenase Increased (Investigations) | 4
Blood Thyroid Stimulating Hormone Increased (Investigations) | 3
High Density Lipoprotein Decreased (Investigations) | 4
White Blood Cell Count Increased (Investigations) | 3
Blood Alkaline Phosphatase Increased (Investigations) | 3
Blood Glucose Increased (Investigations) | 3
Blood Pressure Increased (Investigations) | 1
Glucose Urine Present (Investigations) | 1
High Density Lipoprotein Increased (Investigations) | 3
Protein Urine Present (Investigations) | 1
Bilirubin Conjugated Increased (Investigations) | 2
Blood Bicarbonate Decreased (Investigations) | 2
Blood Insulin Increased (Investigations) | 2
Blood Uric Acid Increased (Investigations) | 2
Sars-Cov-2 Test Positive (Investigations) | 2
Weight Increased (Investigations) | 2
Blood Bicarbonate Increased (Investigations) | 1
Blood Calcium Decreased (Investigations) | 1
Blood Creatine Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Blood Iron Decreased (Investigations) | 1
Blood Magnesium Decreased (Investigations) | 1
Blood Oestrogen Decreased (Investigations) | 1
Blood Phosphorus Decreased (Investigations) | 1
Blood Potassium Decreased (Investigations) | 1
Blood Testosterone Increased (Investigations) | 1
Blood Urea Increased (Investigations) | 1
Blood Urine Present (Investigations) | 1
Chest X-Ray Abnormal (Investigations) | 1
Crystal Urine Present (Investigations) | 1
Electrocardiogram Qt Prolonged (Investigations) | 1
Haematocrit Decreased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 1
Irregular Heart Rate (Investigations) | 1
Leptin Level Increased (Investigations) | 1
Liver Function Test Increased (Investigations) | 1
Mammogram Abnormal (Investigations) | 1
Muscle Strength Abnormal (Investigations) | 1
Neutrophil Count Increased (Investigations) | 1
Pregnancy Test Urine Positive (Investigations) | 1
Red Blood Cells Urine (Investigations) | 1
Transaminases Increased (Investigations) | 1
Urinary Casts (Investigations) | 1
Urine Uric Acid Increased (Investigations) | 1
Weight Decreased (Investigations) | 1
White Blood Cells Urine (Investigations) | 1
White Blood Cells Urine Positive (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 20
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 16
Back Pain (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Neck Pain (Musculoskeletal and connective tissue disorders) | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 2
Morphoea (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Discoid Meniscus (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Greater Trochanteric Pain Syndrome (Musculoskeletal and connective tissue disorders) | 1
Growing Pains (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Joint Hyperextension (Musculoskeletal and connective tissue disorders) | 1
Joint Instability (Musculoskeletal and connective tissue disorders) | 1
Ligament Pain (Musculoskeletal and connective tissue disorders) | 1
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Perthes Disease (Musculoskeletal and connective tissue disorders) | 1
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Immunisation Reaction (Injury, poisoning and procedural complications) | 11
Fall (Injury, poisoning and procedural complications) | 10
Contusion (Injury, poisoning and procedural complications) | 7
Ligament Sprain (Injury, poisoning and procedural complications) | 7
Foot Fracture (Injury, poisoning and procedural complications) | 6
Procedural Pain (Injury, poisoning and procedural complications) | 4
Skin Laceration (Injury, poisoning and procedural complications) | 5
Thermal Burn (Injury, poisoning and procedural complications) | 5
Concussion (Injury, poisoning and procedural complications) | 3
Muscle Strain (Injury, poisoning and procedural complications) | 4
Skin Abrasion (Injury, poisoning and procedural complications) | 3
Joint Dislocation (Injury, poisoning and procedural complications) | 2
Joint Injury (Injury, poisoning and procedural complications) | 3
Wound (Injury, poisoning and procedural complications) | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 2
Limb Injury (Injury, poisoning and procedural complications) | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 2
Post Procedural Fever (Injury, poisoning and procedural complications) | 1
Radius Fracture (Injury, poisoning and procedural complications) | 2
Scar (Injury, poisoning and procedural complications) | 2
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2
Accidental Overdose (Injury, poisoning and procedural complications) | 1
Anaesthetic Complication Vascular (Injury, poisoning and procedural complications) | 1
Animal Scratch (Injury, poisoning and procedural complications) | 1
Bone Fragmentation (Injury, poisoning and procedural complications) | 1
Craniofacial Fracture (Injury, poisoning and procedural complications) | 1
Gingival Injury (Injury, poisoning and procedural complications) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Human Bite (Injury, poisoning and procedural complications) | 1
Incision Site Rash (Injury, poisoning and procedural complications) | 1
Lip Injury (Injury, poisoning and procedural complications) | 1
Nerve Injury (Injury, poisoning and procedural complications) | 1
Sunburn (Injury, poisoning and procedural complications) | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Tongue Injury (Injury, poisoning and procedural complications) | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1
Ulna Fracture (Injury, poisoning and procedural complications) | 1
Anxiety (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 10
Depressed Mood (Psychiatric disorders) | 9
Suicidal Ideation (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 7
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 4
Libido Decreased (Psychiatric disorders) | 4
Libido Increased (Psychiatric disorders) | 4
Panic Attack (Psychiatric disorders) | 4
Stress (Psychiatric disorders) | 2
Mood Altered (Psychiatric disorders) | 3
Obsessive-Compulsive Disorder (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Depressive Symptom (Psychiatric disorders) | 2
Intentional Self-Injury (Psychiatric disorders) | 2
Adjustment Disorder (Psychiatric disorders) | 1
Binge Eating (Psychiatric disorders) | 1
Disturbance In Sexual Arousal (Psychiatric disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Dyssomnia (Psychiatric disorders) | 1
Eating Disorder (Psychiatric disorders) | 1
Emotional Disorder (Psychiatric disorders) | 1
Negativism (Psychiatric disorders) | 1
Sleep Disorder (Psychiatric disorders) | 1
Tension (Psychiatric disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea At Rest (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Crusting (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 41
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Conjunctival Primary Acquired Melanosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign Neoplasm Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 7
Erection Increased (Reproductive system and breast disorders) | 8
Menstruation Irregular (Reproductive system and breast disorders) | 5
Amenorrhoea (Reproductive system and breast disorders) | 3
Spontaneous Penile Erection (Reproductive system and breast disorders) | 4
Breast Cyst (Reproductive system and breast disorders) | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 2
Spontaneous Ejaculation (Reproductive system and breast disorders) | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 2
Uterine Polyp (Reproductive system and breast disorders) | 2
Bartholin's Cyst (Reproductive system and breast disorders) | 1
Breast Fibrosis (Reproductive system and breast disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Breast Swelling (Reproductive system and breast disorders) | 1
Breast Tenderness (Reproductive system and breast disorders) | 1
Dyspareunia (Reproductive system and breast disorders) | 1
Ejaculation Disorder (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Epididymal Cyst (Reproductive system and breast disorders) | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1
Genital Cyst (Reproductive system and breast disorders) | 1
Genital Discomfort (Reproductive system and breast disorders) | 1
Genital Hyperaesthesia (Reproductive system and breast disorders) | 1
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1
Intermenstrual Bleeding (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menstrual Discomfort (Reproductive system and breast disorders) | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1
Painful Erection (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Penile Plaque (Reproductive system and breast disorders) | 1
Polymenorrhoea (Reproductive system and breast disorders) | 1
Premenstrual Pain (Reproductive system and breast disorders) | 1
Testicular Torsion (Reproductive system and breast disorders) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
Vulva Cyst (Reproductive system and breast disorders) | 1
Vulval Disorder (Reproductive system and breast disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5
Vitamin D Deficiency (Metabolism and nutrition disorders) | 6
Dyslipidaemia (Metabolism and nutrition disorders) | 5
Increased Appetite (Metabolism and nutrition disorders) | 5
Appetite Disorder (Metabolism and nutrition disorders) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 4
Folate Deficiency (Metabolism and nutrition disorders) | 4
Iron Deficiency (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperphagia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Lipoedema (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 1
Dry Eye (Eye disorders) | 3
Cataract (Eye disorders) | 3
Eye Pain (Eye disorders) | 3
Corneal Pigmentation (Eye disorders) | 2
Eye Irritation (Eye disorders) | 2
Myopia (Eye disorders) | 1
Scleral Pigmentation (Eye disorders) | 2
Blepharospasm (Eye disorders) | 1
Blindness (Eye disorders) | 1
Conjunctival Haemorrhage (Eye disorders) | 1
Conjunctival Pigmentation (Eye disorders) | 1
Conjunctivitis Allergic (Eye disorders) | 1
Eye Pruritus (Eye disorders) | 1
Eyelid Exfoliation (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Macular Pigmentary Changes (Eye disorders) | 1
Meibomian Gland Dysfunction (Eye disorders) | 1
Retinopathy (Eye disorders) | 1
Swelling Of Eyelid (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Visual Acuity Reduced (Eye disorders) | 1
Visual Impairment (Eye disorders) | 1
Vitreous Degeneration (Eye disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 7
Vertigo (Ear and labyrinth disorders) | 6
Hyperacusis (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Ear Discomfort (Ear and labyrinth disorders) | 1
Ear Disorder (Ear and labyrinth disorders) | 1
Excessive Cerumen Production (Ear and labyrinth disorders) | 1
Inner Ear Inflammation (Ear and labyrinth disorders) | 1
Middle Ear Effusion (Ear and labyrinth disorders) | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1
Vertigo Positional (Ear and labyrinth disorders) | 1
Bladder Pain (Renal and urinary disorders) | 2
Microalbuminuria (Renal and urinary disorders) | 3
Polyuria (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Albuminuria (Renal and urinary disorders) | 1
Calculus Bladder (Renal and urinary disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Glomerulonephritis Membranoproliferative (Renal and urinary disorders) | 1
Glycosuria (Renal and urinary disorders) | 1
Lower Urinary Tract Symptoms (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal Impairment (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Eosinophilia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Scalp Haematoma (Vascular disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Hepatic Steatosis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Liver Opacity (Hepatobiliary disorders) | 1
Metabolic Dysfunction-Associated Liver Disease (Hepatobiliary disorders) | 1
Ocular Icterus (Hepatobiliary disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Sinus Tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Hypertrophy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Adrenal Insufficiency (Endocrine disorders) | 1
Adrenocortical Insufficiency Acute (Endocrine disorders) | 1
Adrenomegaly (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Polycystic Ovarian Syndrome (Endocrine disorders) | 1
Precocious Puberty (Endocrine disorders) | 1
Thyroid Stimulating Hormone Deficiency (Endocrine disorders) | 1
Food Allergy (Immune system disorders) | 2
Seasonal Allergy (Immune system disorders) | 2
Drug Hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Retinitis Pigmentosa (Congenital, familial and genetic disorders) | 2
Hamartoma (Congenital, familial and genetic disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 3
Skin Plaque (Skin and subcutaneous tissue disorders) | 3
Solar lentingo (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information regarding setmelanotide supplied by Rhythm to the investigator is privileged and confidential information. The investigator agrees to use this information to accomplish the study and will not use it for other purposes without consent from Rhythm. The information obtained from the clinical study will be used towards the development of setmelanotide and may be disclosed to regulatory authority(ies), other investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03651765/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03651765/SAP_001.pdf